CLINICAL TRIAL: NCT02966353
Title: A Multicenter Phase II, Open Label, Single Arm Study to Evaluate the Efficacy and Safety of Ruxolitinib in the Treatment of Anemic Myelofibrosis Patients.
Brief Title: Efficacy and Safety of Ruxolitinib in the Treatment of Anemic Myelofibrosis Patients.
Acronym: REALISE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CINC424A2411
Record Dates: First submitted 2016-10-18; First posted 2016-11-17 (Estimated); Results first posted 2020-04-30 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Primary Myelofibrosis; Post-Polycythemia Vera-Myelofibrosis; Post-Essential Thrombocythemia Myelofibrosis
Keywords: Ruxolitinib; anemia; Primary Myelofibrosis; PMF; Post-Polycythemia Vera-Myelofibrosis; PPV-MF; Post-Essential Thrombocythemia Myelofibrosis; PET-MF; adult; INC424
MeSH Terms: conditions — Primary Myelofibrosis; Anemia | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All Subjects (Experimental): 10 mg BID (2 tablets of 5mg) was self-administered as starting dose for all patients. This dose was maintained for the first 12 weeks and titrated up thereafter unless they had met criteria for dose hold or dose reduction. Dose was to have been increased or decreased per standardized dosing paradigm and not to have exceeded 25 mg bid.
  Interventions: Drug: ruxolitinib

INTERVENTIONS:
Drug: ruxolitinib — Ruxolitinib was supplied in 5 mg tablets to be taken orally approximately 12 hours apart (morning and night)

SUMMARY:
This was a study of treatment with ruxolitinib in patients who presented with transfusion dependent or independent anemia. Starting dose was 10 mg BID. This dose was maintained for the first 12 weeks of the study and up-titrated thereafter unless the subject met criteria for dose hold or dose reduction

DETAILED DESCRIPTION:
This was a study of treatment with ruxolitinib in patients who present with transfusion dependent or independent anemia at screening defined as an hemoglobin <10 g/dL with 10 mg BID starting dose with subsequent up titrations (maximum dose 25 mg BID) depending on safety and efficacy. This dosing approach for anemic MF patients will be systematically studied in this prospective multicenter phase II open label single arm trial to determine if the levels of spleen length reduction and symptom improvement are consistent with those reported in previous clinical trials with ruxolitinib in patients with anemia and doses according to platelet counts at the moment of treatment initiation, and whether this lower starting dose and up titration approach may minimize the initial hemoglobin and platelet declines and transfusion requirements.

ELIGIBILITY:
Inclusion Criteria:

Written informed consent must be obtained prior to any screening procedures.

1. Male or female patients aged ≥ 18 years of age.
2. Patients must have been diagnosed with PMF, according to the 2016 revised International Standard Criteria, PPV MF or PET-MF, irrespective of JAK2 mutation status.
3. Patients must have had palpable splenomegaly that is equal to or greater than 5 cm below the left costal margin.
4. Patients must have had hemoglobin less than 10 g/dL
5. Patients must have had a history of transfusions must have a documented transfusion record in the previous 12 weeks to baseline.
6. Patients must have had ECOG performance status of 0, 1, or 2.
7. Patients must have had a peripheral blood blast percentage count of < 10%.
8. Patients must have recovered or stabilized sufficiently from any adverse drug reactions associated with prior treatments before beginning treatment with ruxolitinib.

Exclusion Criteria:

1. Patients who had prior treatment with any JAK1 or JAK2 inhibitor.
2. Patients who had known hypersensitivity to ruxolitinib or other JAK1/JAK2 inhibitors, or to their excipients.
3. Patients who had been eligible for hematopoietic stem cell transplantation (suitable candidate and a suitable donor is available).
4. Patients who had inadequate bone marrow reserve at baseline as demonstrated by at least one of the following:

   1. ANC that is ≤ 1,000/µL.
   2. Platelet count that is <50,000/µL without the assistance of growth factors, thrombopoietic factors or platelet transfusions.
   3. Hemoglobin count that is ≤ 6.5 g/dL despite transfusions.
5. Patients who had severely impaired renal function defined by: Creatinine clearance less than 30 mL/min.
6. Patients who had inadequate liver function defined by any of these:

   1. Total bilirubin ≥ 2.5 x ULN and subsequent determination of direct bilirubin ≥ 2.5 x ULN;
   2. Alanine aminotransferase (ALT) > 2.5 x ULN;
   3. Aspartate aminotransferase (AST) > 2.5 x ULN.
7. Patients who were being treated concurrently with a strong (potent) systemic inhibitor or inducer of CYP3A4 at the time of Screening.
8. Presence of active bacterial, fungal, parasitic, or viral infection which requires therapy.
9. Known history of human immunodeficiency virus (HIV) infection or other immunodeficiency syndromes such as X-linked agammaglobulinemia and common variable immune deficiency.
10. Acute viral hepatitis or active chronic hepatitis B or C infection. Patients with inactive chronic infection (without viral replication) can be enrolled
11. History of progressive multifocal leuko-encephalopathy.
12. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of ruxolitinib .
13. History or current diagnosis of uncontrolled or significant cardiac disease, including any of the following:

    1. Myocardial infarction within last 6 months
    2. Uncontrolled congestive heart failure
    3. Unstable angina within last 6 months
    4. Clinically significant (symptomatic) cardiac arrhythmias (e.g. bradyarrhythmias, sustained ventricular tachycardia, and clinically significant second or third degree AV block without a pacemaker)
14. Significant concurrent, uncontrolled medical condition which, in the investigator's opinion, would have jeopardized the safety of the patient or compliance with the protocol.
15. Patients who were undergoing treatment with another investigational medication or had been treated with an investigational medication within 30 days or 5 half-lives (whichever is longer) prior to the first dose of study drug.
16. Patients who had a history of malignancy in the past 3 years, except for treated early stage squamous or basal cell carcinoma.
17. Patients who were unable to comprehend or are unwilling to sign an ICF.
18. Pregnant or nursing (lactating) women
19. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they were using highly effective methods of contraception throughout the study duration inclusive of 30 day safety follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2018-07-24 (Actual); Study Completion 2019-02-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- Novartis Investigative Site, Vienna, Austria
- Belgium (2):
  - Novartis Investigative Site, Antwerp
  - Novartis Investigative Site, Leuven
- Novartis Investigative Site, Sofia, Bulgaria
- Novartis Investigative Site, Vancouver, British Columbia, Canada
- Novartis Investigative Site, Halle S, Germany
- Novartis Investigative Site, Athens, GR, Greece
- Italy (3):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Palermo, PA
- Novartis Investigative Site, Bunkyo Ku, Tokyo, Japan
- Russia (2):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Petrozavodsk
- Spain (3):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Alicante, Valencia
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Kocaeli

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Screening evaluations were performed to determine the eligibility for the study and establish a baseline prior to dosing.
Period: Overall Study
Arm/Group | All Subjects
Started | 51
Completed After Data Cutoff (One patient completed one week after 30 days follow up for safety) | 1
Completed (Primary reason for discontinuation is presented for reason not completed.) | 29
Not Completed | 22
Not completed — Withdrawal by Subject | 7
Not completed — Adverse Event | 4
Not completed — Death | 4
Not completed — Physician Decision | 3
Not completed — Progressive disease | 2
Not completed — Protocol deviation | 2

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects
Number analyzed (Participants) | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 30
Race/Ethnicity, Customized [Number; unit: participants]
  White | 48
  Asian | 3
Type of myelofibrosis [Number; unit: participants] — Adult Primary Myelofibrosis (PMF): Presence of megakaryocytic proliferation and atypia, accompanied by reticulin and/or collagen fibrosis grades 2 or 3, Post-Polycythemia Vera-Myelofibrosis (PPV-MF): previous diagnosis of polycythemia vera as defined by WHO criteria (Tefferi 2007b) AND Bone marrow fibrosis grade 2-3 (on 0-3 scale)3 or grade 3-4 (on 0-4 scale )4, or Post-Essential Thrombocythemia Myelofibrosis (PET-MF): Documentation of a previous diagnosis of essential thrombocythemia as defined by WHO criteria and bone marrow fibrosis grade 2-3 (on 0-3 scale)3 or grade 3-4 (on 0-4 scale)
  participants
    Primary myelofibrosis | 34
    Post-polycythemia vera myelofibrosis | 6
    Post-essential thrombocythemia myelofibrosis | 11
Time since intial diagnosis [Mean (Standard Deviation); unit: months] | 32.9 (44.16)
Bone Marrow Fibrosis Grade at Diagnosis [Number; unit: participants] — Grades: 0=Scattered linear reticulin with no intersections (cross-overs) corresponding to normal BM, 1=Loose network of reticulin with many intersections, especially in perivascular areas, 2=Diffuse and dense increase in reticulin with extensive intersections, occasionally with focal bundles of thick fibers mostly consistent with collagen, and/or focal, 3=Diffuse and dense increase in reticulin with extensive intersections and coarse bundles of thick fibers consistent with collagen, usually associated with osteosclerosis. Higher grades indicate more fibrosis
  participants
    Grade 0 | 0
    Grade 1 | 6
    Grade 2 | 26
    Grade 3 | 18
    Missing | 1
Constitutional symptoms [Number; unit: participants] — Debilitating constitutional symptoms that include fatigue, weight loss, pruritus, night sweats, fever, and bone, muscle, or abdominal pain
  participants
    Present | 29
    Absent | 22
Palpable spleen length (cm) below costal margin [Mean (Standard Deviation); unit: centimeters] | 11.7 (6.20)
Hemoglobin level [Mean (Standard Deviation); unit: g/dL] | 88.6 (9.74)
Platelets [Mean (Standard Deviation); unit: 10E9/L] | 236.7 (176.88)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least 50% Reduction in Spleen Length From Baseline at Week 24
Description: Percentage of participants achieving a 50% reduction in spleen length at week 24. For subjects with palpable spleen at baseline and non-palpable at post-baseline, the post-baseline spleen are imputed as 0. Subjects who had palpable, but missing spleen length at baseline is excluded from the analysis. Subjects with missing spleen length at Week 24 or who withdraw earlier from the study are considered as a non-responder. The 95% CI is computed using exact Clopper-Pearson method.
Time Frame: Baseline up to week 24
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Subjects
Number analyzed (Participants) | 50
percentage of participants | 56.0 [41.3 to 70.0]

2. Secondary Outcome: Percentage of Participants With at Least 50% Reduction in Spleen Length From Baseline at Week 48
Description: Percentage of participants achieving a 50% reduction in spleen length at week 48. For subjects with palpable spleen at baseline and non-palpable at post-baseline, the post-baseline spleen is imputed as 0. Subjects who had palpable, but missing spleen length at baseline is excluded from the analysis. Subjects with missing spleen length at Week 48 or who withdraw earlier from the study are considered as a non-responder. The 95% CI is computed using exact Clopper-Pearson method.
Time Frame: Baseline up to week 48
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Subjects
Number analyzed (Participants) | 50
percentage of participants | 36.0 [22.9 to 50.8]

3. Secondary Outcome: Percentage of Participants by Spleen Length Reduction or no Increase From Baseline Category at Week 24 and Week 48
Description: Participants who achieved a ≤ 50% reduction in spleen length at week 24 and 48 (reduction) and participants who had no increase greater than or equal to 50% (increase). The edge of the spleen shall be determined by palpation, measured in centimeters, using a soft ruler, from the costal margin to the point of greatest splenic protrusion. For subjects with palpable spleen at baseline and non-palpable at post-baseline, the post-baseline spleen is imputed as 0.
Time Frame: baseline, weeks 24 and 48
Population: Full analysis set n: participants with a value at both Baseline and that time point.
Measure: Number; unit: percentage of participants
Arm/Group | All Subjects
Number analyzed (Participants) | 51
percentage of participants
  Wk 24 ≤ -50% reduction n=43: number analyzed (Participants) | 43
  Wk 24 ≤ -50% reduction n=43 | 65.1
  Wk 24 -50%, -25% reduction n=43: number analyzed (Participants) | 43
  Wk 24 -50%, -25% reduction n=43 | 11.6
  Wk 24 -25%, -5% reduction n=43: number analyzed (Participants) | 43
  Wk 24 -25%, -5% reduction n=43 | 9.3
  Wk 24 -5%, 5% reduction, increase n=43: number analyzed (Participants) | 43
  Wk 24 -5%, 5% reduction, increase n=43 | 4.7
  Wk 24 5%, 25% increase n=43: number analyzed (Participants) | 43
  Wk 24 5%, 25% increase n=43 | 9.3
  Wk 24 25%, 50% increase n=43: number analyzed (Participants) | 43
  Wk 24 25%, 50% increase n=43 | 0
  Wk 24 >50% increase n=43: number analyzed (Participants) | 43
  Wk 24 >50% increase n=43 | 0
  Wk 24 remained non-palpable n=43: number analyzed (Participants) | 43
  Wk 24 remained non-palpable n=43 | 0
  Wk 24 became palpable n=43: number analyzed (Participants) | 43
  Wk 24 became palpable n=43 | 0
  Wk 48 ≤ -50% reduction n=36: number analyzed (Participants) | 36
  Wk 48 ≤ -50% reduction n=36 | 50.0
  Wk 48 -50%, -25% reduction n=36: number analyzed (Participants) | 36
  Wk 48 -50%, -25% reduction n=36 | 22.2
  Wk 48 -25%, -5% reduction n=36: number analyzed (Participants) | 36
  Wk 48 -25%, -5% reduction n=36 | 16.7
  Wk 48 -5%, 5% reduction, increase n=36: number analyzed (Participants) | 36
  Wk 48 -5%, 5% reduction, increase n=36 | 5.6
  Wk 48 5%, 25% increase n=36: number analyzed (Participants) | 36
  Wk 48 5%, 25% increase n=36 | 2.8
  Wk 48 25%, 50% increase n=36: number analyzed (Participants) | 36
  Wk 48 25%, 50% increase n=36 | 2.8
  Wk 48 >50% increase n=36: number analyzed (Participants) | 36
  Wk 48 >50% increase n=36 | 0
  Wk 48 remained non-palpable n=36: number analyzed (Participants) | 36
  Wk 48 remained non-palpable n=36 | 0
  Wk 48 became palpable n=36: number analyzed (Participants) | 36
  Wk 48 became palpable n=36 | 0

4. Secondary Outcome: Percentage of Participants With at Least a 50% Reduction in Myelofibrosis 7 Item Symptom Scale (MF-7) and Myelofibrosis Symptom Assessment Form (MFSAF) at Week 24
Description: The MF-7 is a disease specific questionnaire comprised of 7 items that measures the severity of seven of the most prevalent associated symptoms including: tiredness, early satiety, abdominal discomfort, night sweats, itching (pruritus), bone pain (diffuse not joint or arthritis) and pain under ribs on left side. Each item was scored on a scale ranging from 0 (absent) to 10 (worst imaginable). The MF-7 score is computed as the sum of the observed scores in the individual items to achieve a 0 to 70 score. There would be one recall period of 24 hours used in this questionnaire. A separate question on Inactivity was to be measured for severity of this symptom on a scale from 0 (absent) to 10 (worst imaginable). This would allow the computation of the MFSAF v2.0 questionnaire results, as 6 out of 7 items in the latter PRO are in overlap with MF7 (they also share same 0-10 range Likert scale and ascending order, absent to worst imaginable).
Time Frame: Baseline and week 24
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Subjects
Number analyzed (Participants) | 45
percentage of participants
  MF-7 Total Symptom score | 51.1 [35.8 to 66.3]
  Modified MFSAF v2.0 Total symptom score | 55.6 [40.0 to 70.4]

5. Secondary Outcome: Patient Global Impression of Change (PGIC) at Week 24 and Week 48
Description: The PGIC is comprised of a single question intended to measure a subject's perspective of improvement or deterioration over time relative to treatment. The PGIC uses a seven-point scale where '1' equals very much improved and '7' equals very much worse.
Time Frame: Baseline up to week 48
Population: Participants with PGIC response at that time point
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 51
Participants
  Week 24 n=41 Very much improved: number analyzed (Participants) | 41
  Week 24 n=41 Very much improved | 5
  Week 24 n=41 Much improved: number analyzed (Participants) | 41
  Week 24 n=41 Much improved | 20
  Week 24 n=41 Minimally improved: number analyzed (Participants) | 41
  Week 24 n=41 Minimally improved | 9
  Week 24 n=41 No change: number analyzed (Participants) | 41
  Week 24 n=41 No change | 6
  Week 24 n=41 Minimally worse: number analyzed (Participants) | 41
  Week 24 n=41 Minimally worse | 1
  Week 24 n=41 Much worse: number analyzed (Participants) | 41
  Week 24 n=41 Much worse | 0
  Week 24 n=41 Very much worse: number analyzed (Participants) | 41
  Week 24 n=41 Very much worse | 0
  Week 48 n=33 Very much improved: number analyzed (Participants) | 33
  Week 48 n=33 Very much improved | 5
  Week 48 n=33 Much improved: number analyzed (Participants) | 33
  Week 48 n=33 Much improved | 15
  Week 48 n=33 Minimally improved: number analyzed (Participants) | 33
  Week 48 n=33 Minimally improved | 9
  Week 48 n=33 No change: number analyzed (Participants) | 33
  Week 48 n=33 No change | 4
  Week 48 n=33 Minimally worse: number analyzed (Participants) | 33
  Week 48 n=33 Minimally worse | 0
  Week 48 n=33 Much worse: number analyzed (Participants) | 33
  Week 48 n=33 Much worse | 0
  Week 48 n=33 Very much worse: number analyzed (Participants) | 33
  Week 48 n=33 Very much worse | 0

6. Secondary Outcome: Percentage of Participants Transfusion Independency From Baseline up to Week 96
Description: Percentage is based on number of subjects who are transfusion dependent at baseline. Transfusion dependence (TD) is defined as subjects receiving 6 or more units of transfusions 12 weeks prior to baseline. Transfusion independence (TI) rate is defined as subjects who are transfusion dependent at baseline and require no unit of transfusion for ≥ 12 weeks at any time during the study.
  Transfusion response rate is defined as subjects who are TD at baseline and have 5 or less units of transfusion for ≥ 12 weeks at any time during the study.
Time Frame: Baseline up to week 96
Population: Number of participants that were transfusion dependent at baseline
Measure: Number; unit: percentage of participants
Arm/Group | All Subjects
Number analyzed (Participants) | 9
percentage of participants
  Week 24 transfusion independent rate | 0
  Week 24 transfusion responder rate | 44.4
  Week 48 transfusion independent rate | 0
  Week 48 transfusion responder rate | 66.7
  Week 72 transfusion independent rate | 0
  Week 72 transfusion responder rate | 66.7
  Week 96 transfusion independent rate | 0
  Week 96 transfusion responder rate | 66.7

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 30 days post treatment, up to maximum duration of 100 weeks
Description: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment
Groups:
- All Patients: 10 mg BID (2 tablets of 5mg) was self-administered as starting dose for all patients. This dose was maintained for the first 12 weeks and titrated up thereafter unless they had met criteria for dose hold or dose reduction. Dose was to have been increased or decreased per standardized dosing paradigm and not to have exceeded 25 mg bid.
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 7/51
Serious Adverse Events (participants affected / at risk) | 17/51
Other Adverse Events (participants affected / at risk) | 40/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=51)
Anaemia (Blood and lymphatic system disorders) | 3
Haemolytic anaemia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Aortic valve disease (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 2
Cardiac failure acute (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Crohn's disease (Gastrointestinal disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Bronchitis (Infections and infestations) | 1
Escherichia sepsis (Infections and infestations) | 1
Escherichia urinary tract infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Lower respiratory tract infection bacterial (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Respiratory syncytial virus bronchitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Staphylococcal bacteraemia (Infections and infestations) | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic encephalopathy (Nervous system disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=51)
Anaemia (Blood and lymphatic system disorders) | 17
Thrombocytopenia (Blood and lymphatic system disorders) | 14
Abdominal pain (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 6
Asthenia (General disorders) | 6
Fatigue (General disorders) | 5
Oedema peripheral (General disorders) | 3
Pyrexia (General disorders) | 4
Bronchitis (Infections and infestations) | 3
Oral herpes (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 5
Alanine aminotransferase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 5
Blood alkaline phosphatase increased (Investigations) | 3
Blood creatinine increased (Investigations) | 3
Gamma-glutamyltransferase increased (Investigations) | 6
Platelet count decreased (Investigations) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3
Acute kidney injury (Renal and urinary disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 4
Haematoma (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-03-12): https://cdn.clinicaltrials.gov/large-docs/53/NCT02966353/SAP_000.pdf
  • Study Protocol (2016-09-12): https://cdn.clinicaltrials.gov/large-docs/53/NCT02966353/Prot_001.pdf